CLINICAL TRIAL: NCT02885012
Title: A Safety and Clinical Efficacy Study Measuring Echocardiographic Composite Comparing Ambrisentan (Letairis®) After a Switch From Bosentan (Tracleer®) or Macintentan (Opsumit®) in Treatment of Pulmonary Arterial Hypertension (PAH)
Brief Title: Crossover Study From Macitentan or Bosentan Over to Ambrisentan
Acronym: Letairis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study ending due to lack of enrollment.
Sponsor: Medical University of South Carolina (Other)
Collaborators: Ochsner Health System (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 00046009
Record Dates: First submitted 2016-05-03; First posted 2016-08-31 (Estimated); Results first posted 2019-04-08 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — ambrisentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Switch to Letairis from Bosentan (Experimental): Subjects will be switching treatments from Bosentan (Tracleer) to Ambrisentan (Letairis)
  Interventions: Drug: Ambrisentan
- Switch to Letairis from Macitentan (Experimental): Subjects will be switching treatments from Macitentan (Opsumit) to Ambrisentan (Letairis)
  Interventions: Drug: Ambrisentan

INTERVENTIONS:
Drug: Ambrisentan — At entry to the study following the screen visits, patients will be switched from bosentan to ambrisentan to complete a 24 week trial. The only study intervention will be ambrisentan.
  Other Names: Letairis

SUMMARY:
The purpose of this study is to learn more about the safety and effects of switching treatments from bosentan (Tracleer) or macientan (Opsumit) to ambrisentan (Letairis) over 24 weeks in subjects with Connective Tissue Disease associated Pulmonary Arterial Hypertension (CTD-PAH).

DETAILED DESCRIPTION:
The study will consist of a group of subjects who have been on bosentan for at least three months and a group that has been on macitentan for at least three months. Both groups will be switched to Letairis 5mg daily after the bosentan or macitentan therapy for three months and then increased to a dose of Letairis 10mg daily at week 4 if well tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a Connective Tissue Disease (CTD)
* Age range: 18-80 years old
* Previous Right Heart Catheterization (RHC) demonstrating PAH
* Forced vital capacity (FVC) greater than 50%
* Carbon Monoxide Diffusing Capacity (DLCO) greater than 50%
* World Health Organization (WHO) functional class II or III
* Able to perform a 6 minute walk test (6MWT)
* Stable dose of antihypertensive medications
* Non-pregnant females
* Have to be currently on stable dose of bosentan for at least 3 months
* Adequate acoustic images to allow for transthoracic echocardiography to be performed

Exclusion Criteria:

* Exercise limitation related to a non-cardiopulmonary reason (e.g. arthritis)
* Severe systemic hypertension greater than 170/95
* Patients with a prior history of cardiovascular disease
* WHO functional class IV status
* Patients with severe other organ disease felt by investigators to impact on survival during the course of the study.
* FVC less than 50% of predicted
* DLCO less than 50% of predicted

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-06; Primary Completion 2017-07-07 (Actual); Study Completion 2017-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terrill Huggins, MD, Principal Investigator — Medical University of South Carolina
Locations (2):
- United States (2):
  - Ochsner Medical Center, New Orleans, Louisiana
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Switch to Letairis From Bosentan | Switch to Letairis From Macitentan
Started | 1 | 2
Completed | 1 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Switch to Letairis From Bosentan | Switch to Letairis From Macitentan | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 3
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 53 [NA to NA] — Only one patient in this arm. | 50.5 [44 to 57] | 51.33 [44 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Stroke Volume
Description: Echocardiography is used to estimate the stroke volume, or the amount of blood ejected from the heart with each beat. An average over three beats is used for the estimate and is reported as ml/beat.
Time Frame: Baseline and 24 Weeks
Measure: Mean (Standard Deviation); unit: ml/beat
Arm/Group | Switch to Letairis From Bosentan | Switch to Letairis From Macitentan
Number analyzed (Participants) | 1 | 2
ml/beat | -2.8 (NA) — Only one patient | 8.7 (4.2)

2. Secondary Outcome: Change in EmPHasis-10 Score
Description: Questionnaire-. The questionnaire is designed to determine how pulmonary hypertension affects the patient's life by asking 10 questions which address breathlessness, fatigue, control, and confidence. emPHasis-10 consists of 10 items which address breathlessness, fatigue, control and confidence. Each item is scored on a semantic differential six-point scale (0-5), with contrasting adjectives at each end. A total emPHasis-10 score is derived using simple aggregation of the 10 items. emPHasis-10 scores range from 0 to 50, higher scores indicate worse quality of life.
Time Frame: Baseline and 24 Weeks
Population: Second patient in second arm did not complete questionnaire in week 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Switch to Letairis From Bosentan | Switch to Letairis From Macitentan
Number analyzed (Participants) | 1 | 1
units on a scale | 3 (NA) — Only one patient | 4 (NA) — Only one patient

3. Secondary Outcome: Disease Status as Measured by Change in Biomarker
Description: NT-proBNP Biomarker: BNP is released from cardiac cells in response to increased pressure. The higher the value the worse the disease status.
Time Frame: Baseline and 12 Weeks
Population: Neither subject in group 2 completed week 24 assessment for this outcome so we are reporting changes at week 12 compared to baseline.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Switch to Letairis From Bosentan | Switch to Letairis From Macitentan
Number analyzed (Participants) | 1 | 2
pg/mL | 926 (NA) — only one subject | -78 (362)

ADVERSE EVENTS:
Time Frame: 24 Weeks
Arm/Group | Switch to Letairis From Bosentan | Switch to Letairis From Macitentan
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 1/1 | 0/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Switch to Letairis From Bosentan (N=1) | Switch to Letairis From Macitentan (N=2)
Worsening hypoxemia due to pneumonia treated with a Z-pack (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Mild severity and unrelated to study medication or Study related procedures (MRN 1411151)
Chest pain and worsening PAH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-18): https://cdn.clinicaltrials.gov/large-docs/12/NCT02885012/Prot_SAP_000.pdf